CLINICAL TRIAL: NCT05650801
Title: Effects of Virtual Music Therapy on Burnout Syndrome Among Healthcare Workers in Tertiary Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yanuar Ardani, Principle Investigator, Indonesia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1176
Record Dates: First submitted 2022-11-29; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Burnout, Psychological; Burnout, Professional
MeSH Terms: conditions — Burnout, Psychological; Burnout, Professional | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group 1 (Experimental): Participants who will be given music therapy 3 times a week for 4 weeks in a row. This group will get Maslach Burnout Inventory and Heart Rate Variability score evaluated before and after music therapy intervention.
  Interventions: Other: Music Therapy
- Intervention Group 2 (Experimental): Participants with burnout syndrome who will be given music therapy 5 times a week for 2 weeks in a row. This group will get Maslach Burnout Inventory and Heart Rate Variability score evaluated before and after music therapy intervention.
  Interventions: Other: Music Therapy
- Neutral Group (No Intervention): Participants in this group will not get any music intervention. The maslach burnout inventory and heart rate variability score will be evaluated before and after four weeks without any intervention

INTERVENTIONS:
Other: Music Therapy — Therapy using a traditional music originally from Indonesian culture
  Arms: Intervention Group 1; Intervention Group 2

SUMMARY:
The goal of this clinical trial is to learn about burnout syndrome among healthcare workers in tertiary hospital. The main questions It aims to answer are the effects of music therapy on burnout syndrome among healthcare workers. Participants will get examined using Maslach Burnout Inventory-Human Service Survey and Heart Rate Variability device before and after music therapy intervention.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about burnout syndrome among healthcare workers in tertiary hospital. The main questions It aims to answer are what kind of music therapy used as a non-pharmacological intervention for health workers with Burnout Syndrome, Maslach Burnout Inventory and Heart Rate Variability score in health workers with Burnout Syndrome before and after music therapy, and does music therapy improve Maslach Burnout Inventory and Heart Rate Variability score in health workers with Burnout Syndrome. Participants will get examined using Maslach Burnout Inventory-Human Service Survey and Heart rate variability device before starting the music therapy. Music therapy will be conducted in two groups, one using 3 session a week for 4 weeks and the second group will get 5 session a week for 2 weeks. After all the session are done, participant will get their Maslach burnout inventory and heart rate variability score evaluate. Researchers will compare the results with neutral group without any music therapy to see if there are any positive effects of music therapy to Maslach burnout inventory and heart rate variability score.

ELIGIBILITY:
Inclusion Criteria:

* Agreed to participate in this study by signing an informed consent sheet
* Age above 18 years old
* Working as a healthcare workers at RSUP dr Kariadi and RSUPN dr Cipto Mangunkusuma, these include doctors, nurses, and other supporting healthcare workers

Exclusion Criteria:

* Refuse to participate in this research
* Have chronic diseases such as cancer, thyroid, and cardiovascular disease
* Taking drugs that affect central nervous system
* Hearing loss and disorder
* Psychosis disorder
* Pregnant women
* Does not like music

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-14 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Maslach Burnout Inventory Human Services Survey | 4 weeks
  an instrument developed to capture burnout for health professionals
Heart Rate Variability | 4 weeks
  Heart rate variability (HRV) is the fluctuation in the time intervals between adjacent heartbeats. HRV indexes neurocardiac function and is generated by heart-brain interactions and dynamic non-linear autonomic nervous system (ANS) processes.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN. dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Kacem I, Kahloul M, El Arem S, Ayachi S, Hafsia M, Maoua M, Ben Othmane M, El Maalel O, Hmida W, Bouallague O, Ben Abdessalem K, Naija W, Mrizek N. Effects of music therapy on occupational stress and burn-out risk of operating room staff. Libyan J Med. 2020 Dec;15(1):1768024. doi: 10.1080/19932820.2020.1768024. PMID 32449482